CLINICAL TRIAL: NCT04471454
Title: Verification of the Reliability and Validity of THINC-it Cognitive Test in the Assessment of Cognitive Impairment in Bipolar Depression
Brief Title: Verification of the Reliability and Validity of THINC-it Tool in Bipolar Depression
Status: Completed | Type: Observational
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-03
Record Dates: First submitted 2020-07-12; First posted 2020-07-15 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-08

CONDITIONS: Bipolar Depression
Keywords: Bipolar Depression; cognitive impairment; THINC-it
MeSH Terms: conditions — Bipolar Disorder; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is some cognitive impairment in patients with bipolar depression. THINC-it is a simple, fast and free cognitive assessment tool. It has good reliability and validity in patients with depression, but its application in patients with bipolar depression is not clear. The purpose of this study is to verify the reliability and validity of THINC-it cognitive test in bipolar depression, and to further explore the difference of cognitive impairment between attack and remission of bipolar depression, so as to provide empirical research basis for clinical evaluation-based treatment.

DETAILED DESCRIPTION:
There is some cognitive impairment in patients with bipolar depression. THINC-it is a simple, fast and free cognitive assessment tool. It has good reliability and validity in patients with depression, but its application in patients with bipolar depression is not clear.

This study includes three steps.

1. baseline: demographic data, sequential test THINC-it and standard test tools, clinical scale evaluation, to verify the discriminant validity and parallel validity of THINC-it in bipolar depression.
2. follow-up (1 week): 30-50 patients with stable bipolar depression were evaluated by clinical scale and THINC-it test to verify the test-retest reliability of THINC-it in bipolar depression.
3. follow-up (8 weeks): all patients with bipolar depression were evaluated by clinical scale, THINC-it test, longitudinal comparison data, and the influencing factors of cognitive impairment were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Case group:

  1. Participants in psychiatric outpatients and inpatients are able and willing to provide informed consent.

two。. The participants were male or female aged between 18 and 65, with junior high school education or above.

3. According to DSM-5 criteria, participants were diagnosed with depressive episodes of bipolar disorder.

4. The total score of Young's Mania scale ((YMRS)) of the participants was less than 5.

5. Subjects received stable mood stabilizers at least two weeks before the study visit, such as SSRIs antidepressants.

6. The combination or use of supportive psychotherapy is allowed.

Control group:

1.it did not meet any of the diagnostic criteria of axis I in DSM-5 in the past or at present.

2.18-65 years old, junior high school education or above. 3.have sufficient audio-visual skills to complete the necessary examinations of the study.

4.Willing to participate in this study, and the informed consent form was signed by the subjects.

Exclusion Criteria:

1. Current alcohol and / or substance use disorders.
2. Any drug that may affect cognitive function, such as psychotropic stimulants, corticosteroids, and receptor blockers.
3. Benzodiazepines were used within 12 hours and alcohol consumption within 8 hours before using the THINC-it cognitive test.
4. The patient has some serious physical conditions.
5. The patient received electroconvulsive therapy ((ECT)) in the past 6 months.
6. There are serious negative suicidal concepts and behaviors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Bipolar depression group: samples were collected from outpatients and inpatients of Shanghai Mental Health Center and Shanghai Pudong New area Mental Health Center from January 2020 to December 2020, who met the diagnostic criteria of DSM-5.
  Healthy control group: the sample came from the social recruitment of healthy people who met the criteria of the control group and matched in sex, age and education level. 100 cases were planned to be included in the group.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-07-05 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Composite THINC-it Tool Score | up to 8 week
  The composite THINC-it tool score is the integrated total score of results from performance on five sub-component cognitive tests of the THINC-it tool.
CANTAB reaction time (RTI) | Up to 1 week
  online computer test, RTI evaluates the response speed of movement and psychology, as well as activity time, reaction time, accurate value and error value of response, and calculates the time required to correctly evaluate the occurrence of stimuli in one location.
1-back memory task (1-back) | Up to 1 week
  the subjects' attention, memory, reaction speed and executive function were tested.
Digit Symbol Substitution Test (DSST) | Up to 1 week
  participants in the digital symbol substitution test calculated the correct total number by matching symbols and numbers as soon as possible within 90 seconds according to the coding table.
Trail Making Test B | Up to 1 week
  he subjects calculated the completion time according to the cross-connection of numbers and letters. The higher the score, the more obvious the functional damage.

SECONDARY OUTCOMES:
Sheehan Disability scale (SDS) | Up to 8 week
  Evaluation of the severity of overall functional impairment
HAM-D | Up to 8 week
  Assess the state of depression
HAM-A | Up to 8 week
  Assessing anxiety state

CONTACTS AND LOCATIONS:
Overall Officials: Jun Chen, M.D., Ph.D, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center IRB, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided